CLINICAL TRIAL: NCT01289106
Title: Open-Label, Randomized Controlled Trial Comparing Three Strategies of Hepatitis B Vaccination in HIV-1-Infected Patients With CD4 Cell Counts Above 200 permm3 and Suppressed Viral Load
Brief Title: Modified Dose and Schedule of Recombinant Hepatitis B Vaccination in HIV-infected Adult Subjects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Kanokporn Chaiklang, Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MED-10-10-21A-13
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-01

CONDITIONS: HIV Infection
Keywords: Hepatitis B vaccine; HIV infection; Modified HBV vaccine dose; Modified HBV vaccine schedule
MeSH Terms: conditions — HIV Infections; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator): 20 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1 and 6 months
  Interventions: Biological: Hepavax-Gene
- Arm B (Experimental): 20 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1,2 and 6 months
  Interventions: Biological: Hepavax-Gene
- Arm C (Experimental): 40 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1,2 and 6 months
  Interventions: Biological: Hepavax-Gene

INTERVENTIONS:
Biological: Hepavax-Gene — 20 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1 and 6 months
  Other Names: Berna
  Arms: Arm A
Biological: Hepavax-Gene — 20 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1,2 and 6 months
  Other Names: Berna
  Arms: Arm B
Biological: Hepavax-Gene — 40 μg of Hepavax-gene intramuscularly injections at deltoid region at 0,1,2 and 6 months
  Other Names: Berna
  Arms: Arm C

SUMMARY:
The purposes of this study include 1) to compare the seroconversion rate of an intensive standard-dose regimen (0, 1, 2 and 6 months) to a standard-dose regimen (0,1 and 6 months), and 2) to compare the seroconversion rate of an intensive double-dose regimen (40 μg at 0,1,2 and 6 months) to a standard-dose regimen (20 μg at 0,1 and 6 months) of HBV vaccine in HIV-infected adult patients.

DETAILED DESCRIPTION:
HIV and HBV share similar risk factors and routes of transmission. HIV/HBV coinfection is associated with greater chance of chronic HBV carrier state, higher level of HBV replication and increasing its potential for transmission. Currently, there are no concrete data to determine the best HBV vaccination schedule in HIV-infected patients. Standard HBV vaccination (20 μg at 0, 1 and 6 months) gives seroconversion rate of 33-63% in HIV-infected individuals compared with >90% in healthy individuals. This study aims to compare the efficacy of an intensive standard-dose regimen (0, 1, 2 and 6 months) to a standard-dose regimen (0,1 and 6 months) and to compare the seroconversion rate of an intensive double-dose regimen (40 μg at 0,1,2 and 6 months) to a standard-dose regimen (20 μg at 0,1 and 6 months) of HBV vaccine in HIV-infected adult patients with CD4 level above 200 permm3 and suppressed viral load.

ELIGIBILITY:
Inclusion Criteria:

* Positive for anti-HIV antibody
* At least 18 years of age
* CD4 > 200 cell/mm3
* On antiretroviral therapy
* Viral load < 50 copies/ml
* Negative for any HBV serological marker (HBsAg, Anti-HBs, Anti-HBc)
* No history of previous hepatitis B vaccination
* Anti-HCV negative
* No active opportunistic infection at the time of screening
* Willing to sign informed consent
* Able to follow up

Exclusion Criteria:

* Pregnancy or breast feeding
* History of hypersensitivity to any component of vaccine
* Diagnosis of malignancy and receiving chemotherapy or radiation
* Other immunocompromised conditions not related to HIV infection (solid-organ transplantation, chemotherapy in the last 6 months)
* On Immunosuppressive treatment, immunomodulating treatment or corticosteroid (equal or above 0.5 mg per kg per day of prednisolone)
* Renal failure (creatinine clearance < 30 mL/min)
* Decompensated cirrhosis (child-pugh C)
* Not able to follow up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate (percentage of subjects with anti-HBs antibody titer >= 10 IU/L) at day 210 | Day 210
  1. To compare the seroconversion rate at day 210 of an intensive standard-dose regimen (0, 1, 2 and 6 months) to a standard-dose regimen (0,1 and 6 months)
  2. To compare the seroconversion rate at day 210 of an intensive double-dose regimen (40 μg at 0,1,2 and 6 months) to a standard-dose regimen (20 μg at 0,1 and 6 months) of HBV vaccine in HIV-infected adult patients

SECONDARY OUTCOMES:
Seroprotective rate (percentage of subjects with anti-HBs antibody titer >= 10 IU/L) at 1 year | 1 year
  To determine the seroprotective rate at 1 year of each of the vaccination regimens.
Number of subjects with adverse events after vaccination | 180 days
  Adverse events include pain at injected site, swelling at injected site, redness at injected site, fever, headache, fatique and anaphylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Kanokporn Chaiklang, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

REFERENCES:
- [Derived] Chaiwarith R, Praparattanapan J, Kotarathititum W, Wipasa J, Chaiklang K, Supparatpinyo K. Higher rate of long-term serologic response of four double doses vs. standard doses of hepatitis B vaccination in HIV-infected adults: 4-year follow-up of a randomised controlled trial. AIDS Res Ther. 2019 Nov 11;16(1):33. doi: 10.1186/s12981-019-0249-8. PMID 31711528
- [Derived] Chawansuntati K, Chaiklang K, Chaiwarith R, Praparattanapan J, Supparatpinyo K, Wipasa J. Hepatitis B Vaccination Induced TNF-alpha- and IL-2-Producing T Cell Responses in HIV- Healthy Individuals Higher than in HIV+ Individuals Who Received the Same Vaccination Regimen. J Immunol Res. 2018 Feb 27;2018:8350862. doi: 10.1155/2018/8350862. eCollection 2018. PMID 29682590
- [Derived] Chaiklang K, Wipasa J, Chaiwarith R, Praparattanapan J, Supparatpinyo K. Comparison of immunogenicity and safety of four doses and four double doses vs. standard doses of hepatitis B vaccination in HIV-infected adults: a randomized, controlled trial. PLoS One. 2013 Nov 12;8(11):e80409. doi: 10.1371/journal.pone.0080409. eCollection 2013. PMID 24265819